CLINICAL TRIAL: NCT00651560
Title: Vytorin As Strategy To Reduce Dislipidemia In Adults
Brief Title: Vytorin As Strategy To Reduce Dislipidemia In Adults (0653A-148)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0653A-148; MK0653A-148; 2008_008
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — Ezetimibe, Simvastatin Drug Combination

INTERVENTIONS:
Drug: ezetimibe (+) simvastatin — ezetimibe 10mg (+) simvastatin 20 mg once daily for 4 weeks of treatment.
  Other Names: Vytorin®; MK0653A

SUMMARY:
This study is intended to allow physicians to check the superior clinical efficacy of Vytorin compared to atorvastatin, as the most adequate therapy using the ATP-III goals achievement and cardiovascular risk reduction in adult patients with dislipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients Who Voluntary Accept To Participate In The Study After Been Informed By The Doctor And Signed The Informed Consent Form.

Exclusion Criteria:

* Any Another Kind Of Contraindication For Use Of Statins
* Hypersensitivity To Any Of The Active Ingredients
* Increased Serum Hepatic Enzymes (Over 3 Times Only)
* Patients With Severe Hepatic Insufficiency
* Women who are Pregnant or Potentially Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2005-11-01 (Actual); Primary Completion 2005-12-23 (Actual); Study Completion 2005-12-23 (Actual)

PRIMARY OUTCOMES:
Evaluate the hypolipidemic effect of Vytorin after 4 weeks treatment in adult patients with mix dislipidemia to reduce the cardiovascular risk and achieve the ATP-III goals. | After 4 weeks treatment

SECONDARY OUTCOMES:
To determine the capability of Vytorin to allow adults patients with dislipidemia and previously treated with atorvastatin to get further reduction of the cardiovascular risk and to achieve the ATP-III goals. | After 4 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC